CLINICAL TRIAL: NCT00345111
Title: ACRYSOF® Restor Apodized Diffractive IOL Postmarket Evaluation of Clinical Outcomes and Life-Style Visual Performance With RESTOR IOL Compared With SN60WF IOL (Control Group)
Brief Title: ACRYSOF® Restor Apodized Diffractive IOL Postmarket Evaluation of Clinical Outcomes and Life-Style Visual Performance RESTOR IOL SN60WF IOL (Control Group)
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Verified with former investigator that recruitment activity did not take place
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 062005-060
Record Dates: First submitted 2006-06-23; First posted 2006-06-27 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Refractive Assessment
Keywords: Restor IOL versus Conventional IOL

INTERVENTIONS:
Procedure: Clinical visual outcomes of bilateral implantation of Restore Intra Ocular Lens.

SUMMARY:
The objective of the research on the Restore Intra Ocular Lens Implant (IOL) is to determine the clinical visual outcomes following bilateral implantation of the IOL compared to a control IOL and to demonstrate what percentage of the subjects obtain spectacle freedom.

DETAILED DESCRIPTION:
The Acusof Restor IOL has recently been FDA approved. This research will be an indicator by comparison to a conventional implant lens used for catract surgery. The standard of care for cataract surgery is to implant an IOL to allow the patient distant vision only. As a result, the patient is forced to wear reading glasses or magnifying glasses for near work. With the Restore IOL implant, the patient will have the ability to be corrected for not only distance vision but for near and intermediate visual needs. With FDA approval, the statistical indications demonstate 80% of patients tested in clinical trials did not have the need for use of glasses after cataract surgery. This research will further confirm and quantify the data already submitted by comparing the control group with the Restore Group in this Phase IV project.

The control group of subjects will be patients who have already had cataract surgery in both eyes approximately 6 months prior to entering the study. These individuals will be tested only for the 6 month evaluation in both eyes, including the following tests (manifest refraction, which determines the best vision correction possible, the near, intermediate and distant visual acuity will be assessed at the respective ranges of distance. contrast sensitivity will be determined by choosing the circles that have lines in them opposed to the ones that don't (further assessing visual acuity), stereopsis which indicates whether both eyes are functioning together, pupilometry which measures the pupil diameter, the life style questionaire and the life style vision evaluation form as well.

The Restore IOl group of subjects' post operative visual acuity data will be compared to the control subjects' post operative visual data results at the distance, near, and intermediate ranges, as well as all the other testing required at the sixxth month time frame listed above. The testing will require approximately 2 hours for the 6 month visit for both control and Restore groups.

The Restore group of subjects will have 4 other visits. The pre operative visit will take avout 2 hours and include the following tests: Manifest refraction, near, inermediate, and distance visual acuity testing, life style questionnaire, and obtaining informed consent. The 1 week and 1 month post-operative visit will include manifest refraction, near, intermediate, and distance visual acuity assessment.

ELIGIBILITY:
Inclusion Criteria: 70 years of age or younger; any race; either gender; diagnosis of cataracts both eyes; pre-existing physical conditions that could skew visual results, such as Diabetes, Retinal detachment, Macular degeneration, or Cancer; subjects must have < 1.00 diopter of astigmatism; biometry results for the Restore patients should target emmetropia or +0.25.

-

Exclusion Criteria: Over 70 years old; other procedures needed at the time of surgery besides cataract extraction; Sulcus-Sulcus or Bag-Sulcus fixation during surgery; Capsulothexis edge not covering optic edge 360 degrees around; Capsular Rupture; vitreous loss; capsularhexis tear; significant anterior chamber hyphema; Zonular rupture.

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
manifest refraction, contrast sensitivity, stereopsis.

SECONDARY OUTCOMES:
near, intermediate and distant visual acuity, life style questionaire and the life style vision evaluation

CONTACTS AND LOCATIONS:
Overall Officials: R. Wayne Bowman, M.D., Principal Investigator — University of Texas, Southwestern Medical Center at Dallas
Locations (1):
- University of Texas Southwestern Medical Center at Dallas, Dallas, Texas, United States